CLINICAL TRIAL: NCT01419353
Title: Programming by Estrogen Treatment in Gonadotropin Releasing Hormone Antagonist Protocol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Antagonist_prog
Record Dates: First submitted 2011-08-01; First posted 2011-08-18 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2011-08

CONDITIONS: Infertility
Keywords: Infertility, IVF, Estrogen
MeSH Terms: conditions — Infertility | interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Follicular Estrogen, Antagonist, IVF (Experimental): Follicular Estrogen in Antagonist IVF protocol
  Interventions: Drug: estradiol valerate
- long IVF protocol (Active Comparator): long IVF protocol
  Interventions: Drug: estradiol valerate

INTERVENTIONS:
Drug: estradiol valerate — 2 mg P.O / day for 1-6 days.

SUMMARY:
The purpose of this study is to determine if pretreatment with Estrogen can assist in the planning and programming of In Vitro Fertilization treatments.

DETAILED DESCRIPTION:
A randomised controlled trial in which study group will be given estrogen derivative before ovarian stimulation in GnRH antagonist protocol and compared to the classical GnRH agonist protocol.Estrogen will be given P.O , "PROGYNOVA' , in a dose of 2 mg /d, starting day 2 of menses and until first Monday to follow. Main outcome measure will be ability to control the ovum pickup day, calculated as a rate of ideal pickups divided by the entire pickup number. All women enrolled will be under 38 years of age, with a clear indication for IVF other than ovulatory dysfunction. women with past 4 treatment failures will be excluded as well as cases in which sperm achieved in surgical methods.

ELIGIBILITY:
Inclusion Criteria:

* IVF treatment in the following indications: Male, Mechanical, Unexplained
* Age<38 years
* Treatment Cycle number 1-4

Exclusion Criteria:

* Ovulatory disorder as an indication for IVF
* Repeated failure in previous IVF treatments (> than 4 cycles)
* Sperm used for treatment was retrieved by surgical procedure

Max Age: 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2011-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
ovum pickup rate that took place between Sunday to Thursday without a compromise | a year
  number of Pickups that took place between Sunday to Thursday (without a compromise in treatment) \ by the entire pickup number

SECONDARY OUTCOMES:
pregnancy rate | a year
  comparison of pregnancy rate between the 2 groups. calculated per cycle

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Shulman, MD, Study Chair — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel, Israel

REFERENCES:
- [Derived] Hershko Klement A, Berkovitz A, Wiser A, Gonen O, Amichay K, Cohen I, Ghetler Y, Shulman A. GnRH-antagonist programming versus GnRH agonist protocol: a randomized trial. Eur J Obstet Gynecol Reprod Biol. 2015 Feb;185:170-3. doi: 10.1016/j.ejogrb.2014.12.021. Epub 2014 Dec 29. PMID 25594526